CLINICAL TRIAL: NCT03052699
Title: Medium and Long-term Complications of the Patients Having Had a Vaginal Caesarian in Hospital René Dubos
Acronym: CeVag
Status: Completed | Type: Observational
Sponsor: Hôpital NOVO (Other)
Responsible Party: Sponsor
Other Study IDs: CHRD1115
Record Dates: First submitted 2016-09-13; First posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2017-02

CONDITIONS: Complications; Cesarean Section
Keywords: Complications; Cesarean Section

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- vaginal Cesarean Section: patients operated to vaginal Cesarean Section
  Interventions: Procedure: vaginal Cesarean Section

INTERVENTIONS:
Procedure: vaginal Cesarean Section — follow-up to patients operated for vaginal Cesarean Section

SUMMARY:
This database has for objective to include the medical data of patients which underwent a vaginal Cesarean Section in our establishment. This collection will allow to determine the risk factors of the maternal morbi-mortality and to estimate the long-term results

DETAILED DESCRIPTION:
It is about an operating technique little known which is used as an alternative of the abdominal Cesarean Section for very premature pregnancies and the main indication is the maternal rescue.

It has several advantages: simplicity of the technique, the dissection of tissues is limited, low risk of bleeding and no abdominal scar.

The purpose is to determine the risk factors of the maternal morbi-mortality and to estimate the long-term results

ELIGIBILITY:
Inclusion Criteria:

* patients operated to vaginal Cesarean in Hospital Rene DUBOS

Exclusion Criteria:

* patients followed in a maternity which do not participate to the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients operated to vaginal Cesarean in Hospital Rene DUBOS
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2015-09; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Risk factors of the maternal morbi-mortality by collection of adverse events during the pregnancy, concomitant pathologies and antecedents | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: MARKOU Georges, PH, Principal Investigator — Rene Dubos Hospital

IPD SHARING:
Plan to Share IPD: No